CLINICAL TRIAL: NCT03060473
Title: TREAT: Treatment of ppROM With Erythromycin vs. Azithromycin Trial
Brief Title: Treatment of ppROM With Erythromycin vs. Azithromycin Trial
Acronym: TREAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient population that meets study criteria is insufficient to continue project in a reasonable amount of time. To continue is futile in resources, staff time, and effort.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-0323
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Preterm Premature Rupture of Membranes (PPROM)
Keywords: PPROM; Azithromycin; Erythromycin
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Azithromycin; Erythromycin; Ampicillin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention model: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin (Experimental): Ampicillin 2 gm IV every 6 hours followed by amoxicillin 500 mg PO every 8 hours with Azithromycin 1 gm PO once at randomization.
  Interventions: Drug: Azithromycin; Drug: Ampicillin; Drug: Amoxicillin
- Erythromycin (Active Comparator): Ampicillin 2 gm IV every 6 hours followed by amoxicillin 250 mg PO every 8 hours for 5 days with erythromycin 250 mg IV every 6 hours for 48 hours followed by 500 mg PO every 8 hours for 5 days.
  Interventions: Drug: Erythromycin; Drug: Ampicillin; Drug: Amoxicillin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 1 gm PO once
  Arms: Azithromycin
Drug: Erythromycin — Erythromycin 250 mg IV every 6 hours for 48 hours followed by 500 mg PO every 8 hours for 5 days.
  Arms: Erythromycin
Drug: Ampicillin — Ampicillin 2 gm IV every 6 hours for 2 days
Drug: Amoxicillin — Amoxicillin 500 mg PO every 8 hours for 5 days (Azithromycin ARM) Amoxicillin 250 mg PO every 8 hours for 5 days (Erythromycin ARM)

SUMMARY:
Preterm premature rupture of membranes (PPROM) complicates 4% of pregnancies annually. This pregnancy complication is a major contributor to preterm births and results in neonatal morbidity and mortality. The current standard of care for PPROM subjects between the gestational age of 24 weeks and 0 days and 33 weeks and 6 days, is to administer ampicillin and erythromycin for a total of 7 days. Erythromycin can cause GI upset and some subjects do not tolerate this regimen over the course of 7 days. In addition, there is a national shortage of erythromycin, and published expert opinion proposed to use a second-generation macrolide (azithromycin) instead of erythromycin. Azithromycin can be taken once daily, is cheaper than erythromycin and has less GI upset adverse effects. The investigators' objective is to compare the effectiveness of the 2 regimens in prolonging pregnancy after PPROM. The investigators' working hypothesis is that there is no measurable difference in the primary outcome between the group randomized to the azithromycin regimen versus the group randomized to the erythromycin regimen.

DETAILED DESCRIPTION:
In the United States, preterm premature rupture of membranes (PPROM) complicates 4% of pregnancies annually. This pregnancy complication is a major contributor to preterm births and results in neonatal morbidity and mortality. Without treatment, 70-80% of women deliver within the 1st week following membrane rupture. Multiple trials have proven that antibiotics given to this population prolong the latency from time of PPROM to delivery, hence reducing maternal and neonatal morbidities.

According to the American College of Obstetrics and Gynecology, the current standard of care for PPROM subjects between the gestational age of 24 weeks and 0 days and 33 weeks and 6 days, is to administer ampicillin 2 gm IV every 6 hours for 48 hours followed by amoxicillin 250 mg orally every 8 hours for 5 days, with erythromycin 250 mg IV every 6 hours for 48 hours followed by 500 mg orally every 8 hours for 5 days. In this regimen, multiple doses of intravenous (IV) and oral (PO) doses of erythromycin are needed to achieve the desired outcome. Erythromycin can cause GI upset and some subjects do not tolerate this regimen over the course of 7 days. In addition, there is a national shortage of erythromycin, and published expert opinion proposed to use a second-generation macrolide (azithromycin) instead of erythromycin. This strategy was adopted nationwide including the maternal center at UTMB since 2014. Compared to erythromycin, advantages of azithromycin include:

* It is taken once orally (due to its long intracellular half-life).
* The entire regimen is much cheaper than the multiple does of erythromycin (23 doses).
* It has less gastrointestinal adverse effects.

As a result, azithromycin is now commonly being used as a substitute for erythromycin on many labor and delivery units around the country.

Despite its common use, there exists no level 1 evidence that azithromycin is equivalent to erythromycin. Haas and colleagues published a retrospective comparison of the two regimens in 2014 and concluded that the substitution of azithromycin for erythromycin in the recommended antibiotic regimen did not impact latency or any other measured maternal or fetal outcomes. This study, however, was limited by its non-randomized retrospective nature.

The investigators' objective is to compare the effectiveness of the 2 regimens in prolonging pregnancy after PPROM.

This trial will be a comparative effectiveness pragmatic randomized trial performed in singleton pregnancies with the diagnosis of PPROM between 24 weeks and 0 days - 32 weeks and 6 days. It will be comparing two well-accepted standardized treatments of care in this subject population: Erythromycin (FDA Category B) versus Azithromycin (FDA Category B). The investigators' primary outcome will be the proportion of women still pregnant by day 7 after the diagnosis of PPROM is made. The investigators' working hypothesis is that there is no measurable difference in the primary outcome between the group randomized to the azithromycin regimen versus the group randomized to the erythromycin regimen. The investigators' secondary outcome will be latency defined as interval from PPROM to delivery.

Data to be collected will consist of demographics, obstetrical history, relevant vital signs and laboratories. Examples of data to be collected but not limited to include: age, ethnicity/race, gravida, para, received tocolytics, received antenatal steroids, gestational age at rupture of membranes, reason for delivery, mode of delivery, gestational age at delivery, chorioamnionitis, date & time of initiation of antibiotics, date & time of delivery, placental abruption, hospital length of stay, number of women undelivered at day 7 of admission, NICU admission, infant intubation days, neonatal NEC and neonatal sepsis.

In addition, drug adverse effects profiles between the two will be assessed in a post treatment patient survey. The latter will be assessing the severity and incidence of diarrhea and other symptoms such as nausea and vomiting and their severity.

The investigators propose a total of 324 subjects will be needed to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age ≥ 18 years and <50 years
* Pregnant women between the gestational age 23 6/7 and 32 6/7 weeks
* Singleton pregnancy
* Preterm premature rupture of membranes, determined clinically
* Cervical dilation visually ≤ 5cm on sterile speculum exam.
* Planned delivery at John Sealy Hospital (JSH)

Exclusion Criteria:

* Intrauterine fetal demise (no fetal heart beat identified and documented by two physicians)
* Any contraindication to expectant management (e.g. fetal compromise, chorioamnionitis, placental abruption)
* Cervical cerclage in place
* Placenta previa or other known placental anomalies
* Contraindication to any of the antibiotics used (allergy to macrolides).
* Enrolled in another trial that may affect outcome.
* Clinical chorioamnionitis or any other active bacterial infection (e.g. pyelonephritis, pneumonia, abscess) at time of randomization: because standard antibiotic therapy for these conditions may confound trial intervention.
* No prenatal care (less than 2 prenatal visits)
* Non-resident subject who is unlikely to be followed-up after delivery
* Any fetal congenital anomaly.
* Significant liver disease defined as known cirrhosis or elevated transaminases of at least 3-fold upper limit of normal
* Significant renal disease defined as serum creatinine known to be >2.0 mg/dl or on dialysis.
* Active congestive heart failure (EF<45%) or pulmonary edema.
* Immunosuppressed subjects: i.e., taking systemic immunosuppressants or steroids (e.g. transplant subjects; not including steroids for lung maturity), HIV with CD4<200, or other.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is to be carried out on pregnant patients with diagnosis of PPROM.
Enrollment: 21 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nkechinyere Emezienna, MD, Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - St. David's North Austin Medical Center, Austin, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol was terminated early due to low accrual and deemed futile.
Period: Overall Study
Arm/Group | Azithromycin | Erythromycin
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Erythromycin | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 24.9 [18 to 31] | 27.56 [21 to 38] | 26.16 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 3 | 4
  White | 9 | 7 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women Still Pregnant by Day 7
Description: Proportion of women still pregnant by day 7 after the diagnosis of PPROM is made. The investigators' working hypothesis is that there is no measurable difference in the primary outcome between the group randomized to the azithromycin regimen versus the group randomized to the erythromycin regimen
Time Frame: 7 days
Population: No data collected. The protocol was closed early due to low accrual and deemed futile.
Arm/Group | Azithromycin | Erythromycin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Latency Defined as Interval From PPROM to Delivery.
Description: Number of days from diagnosis of PPROM to delivery
Time Frame: 7 days
Population: No data collected. The protocol was closed early due to low accrual and deemed futile.
Arm/Group | Azithromycin | Erythromycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Azithromycin | Erythromycin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No data collected. The protocol was closed early due to low accrual and deemed futile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03060473/Prot_SAP_000.pdf